CLINICAL TRIAL: NCT01469585
Title: Oral Contraceptives and Subantimicrobial Doxycycline: Effect on Endometrial Matrix Metalloproteinases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Charles Drew University of Medicine and Science (Other); Meharry Medical College (Other)
Responsible Party: Principal Investigator, Bliss Kaneshiro, Assistant Professor, University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UH DOXY RTRN
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Breakthrough Bleeding
Keywords: continuous oral contraceptives; Matrix Metalloproteinase expression
MeSH Terms: conditions — Metrorrhagia | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sub-antimicrobial doxycycline (Active Comparator): Women will take sub-antimicrobial doxycyline in addition to the continuous oral contraceptive pill.
  Interventions: Drug: Doxycycline
- Continuous Oral Contraceptive Pill (No Intervention): Women will take only the continuous oral contraceptive.

INTERVENTIONS:
Drug: Doxycycline — 40 mg orally at the start of cycle 3 (study day 57) for 28 days.
  Other Names: Oracea
  Arms: Sub-antimicrobial doxycycline

SUMMARY:
The purpose of this study is to compare the effects (good and bad) of subantimicrobial dose doxycycline on the irregular bleeding women experience when taking continuous oral contraceptive pills. This research is being done because currently, there is no effective treatment for this condition. Findings from this study could help to decrease the side effects of birth control pills and decrease unplanned pregnancies.

DETAILED DESCRIPTION:
Continuous oral contraceptive administration entails women taking hormonally active pills for 28 days without a seven day placebo week to avoid hormonal withdrawal bleeding. Unfortunately, with continuous administration, timed, regular bleeding can be replace by irregular, unscheduled bleeding, which often leads to dissatisfaction, discontinuation and the possibility of unplanned pregnancy.

Matrix Metalloproteinases, a group of zinc-dependant proteases, are hypothesized to play a role in endometrial degradation. The purpose of this study is to describe the expression of Matrix Metalloproteinases in endometrial biopsy specimens collected 1) prior to initiating oral contraceptives 2) while taking cyclic oral contraceptive 3) while taking continuous oral contraceptives and 4) while taking continuous oral contraceptives along with sub-antimicrobial doxycycline.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages 18 and 45 who are ovulatory as demonstrated by a pre-treatment Progesterone (P) greater than or equal to 3.0 ng/mL prior to oral contraceptive use

Exclusion Criteria:

* Women with any absolute contraindications to ethinyl estradiol and levonorgestrel;
* Women who are pregnant or breastfeeding
* Use of oral contraceptives, patch, ring, intrauterine or implantable hormonal contraception within 4-weeks;
* Medroxyprogesterone acetate use within six months;
* Current use of drugs that interfere with sex steroid metabolism.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bliss Kaneshiro, MD, MPH, Principal Investigator — University of Hawaii John A. Burns School of Medicine Department of Obstetrics and Gynecology
Locations (1):
- Kapiolani Medical Center for Women and Children, Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sub-antimicrobial Doxycycline | Continuous Oral Contraceptive Pill
Started | 11 | 9
Completed | 4 | 6
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Active Comparator: Subantimicrobial Doxycycline: Active comparator: Subantimicrobial doxycycline
- No Intervention: Continuous Oral Contraceptive Pill: No intervention: Continuous oral contraceptive pill
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Subantimicrobial Doxycycline | No Intervention: Continuous Oral Contraceptive Pill | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 2 | 7
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Endometrial Matrix Metalloproteinase Expression by Gel Densitometry
Description: Baseline Matrix Metalloproteinase expression (activity level) will be determined on day 19-21 of cycle 1. During cycle 2, when women are taking the cyclic oral contraceptive, the endometrial biopsy will be performed between cycle day 19-21 (study day 47-49), prior to endometrial degradation and activity level will be noted. Of note, the outcome is MMP activity level, not a change in level.
Time Frame: 49 days
Measure: Mean (Standard Deviation); unit: relative expression
Groups:
- Sub-antimicrobial Doxycycline Group: Sub-antimicrobial doxycycline group (controlled release subantimicrobial doxycycyline 40 mg once daily)
- Control: Control (no medication)
Arm/Group | Sub-antimicrobial Doxycycline Group | Control
Number analyzed (Participants) | 11 | 9
relative expression | 1.33 (0.41) | 2.49 (0.72)

2. Secondary Outcome: Matrix Metalloproteinase Expression and Activity by Gel Densitometry
Description: Based on doxycycline's action as an Matrix Metalloproteinase inhibitor, it is hypothesized that Matrix Metalloproteinase expression and activity level will be decreased in women taking sub-antimicrobial doxycycline compared to women on continuous oral contraceptives only. The outcome is activity level (not a change in activity level)
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: relative expression
Arm/Group | Sub-antimicrobial Doxycycline | Continuous Oral Contraceptive Pill
Number analyzed (Participants) | 4 | 6
relative expression | 1.52 (0.63) | 1.98 (0.87)

ADVERSE EVENTS:
Arm/Group | Sub-antimicrobial Doxycycline | Continuous Oral Contraceptive Pill
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No